CLINICAL TRIAL: NCT00208208
Title: Geodon (Ziprasidone) for Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2001-0261; Grant 2001-0261
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2005-04

CONDITIONS: Posttraumatic Stress Disorder; Post-Traumatic Stress Disorder; PTSD
Keywords: Posttraumatic Stress Disorder; Post-traumatic Stress Disorder; PTSD; Geodon; Ziprasidone
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — ziprasidone

INTERVENTIONS:
Drug: Ziprasidone

SUMMARY:
Atypical antipsychotics have shown promise in the treatment of depression and anxiety, which are prominent symptoms of PTSD. The profile of the atypical antipsychotic, ziprasidone (Geodon), suggests possible anxiolytic and antidepressant properties. This research will assess the potential effectiveness of Geodon in civilian men and women who suffer from severe PTSD. Response to ziprasidone or placebo will be measured by Clinician Administered PTSD Scale (CAPS) and Treatment Outcomes PTSD Scale (TOP-8).

DETAILED DESCRIPTION:
PTSD is a common disorder with 10% lifetime prevalence among Americans. The major causes of PTSD are sexual assault, accidents, disasters Despite this public health burden, only two drugs, sertraline (Zoloft) and paroxetine (Paxil), are approved by the FDA for the treatment of PTSD. New options for the treatment of PTSD are much needed. Approximately half of patients with PTSD respond to Zoloft and Paxil. Many patients experience psychotic symptoms with PTSD, which may not respond to treatment to Zoloft and Paxil.

Though classified as an anxiety disorder in the DSM-IV, PTSD is accompanied by psychotic symptoms in almost half of patients (Butler et al 1996; Hamner et al 1999, Lindley et al 2000). Also, PTSD has an extensive comorbidity with major depressive disorder (Davis et al 2000). While Geodon is approved by the FDA in the United States for the treatment of psychosis, it has not been evaluated for the treatment of PTSD . A clinical trial of Geodon in PTSD will help delineate the potential antidepressant spectrum of efficacy of Geodon as well as its anxiolytic profile.

ELIGIBILITY:
Inclusion Criteria:

* Men & women with DSM-IV clinical diagnosis of PTSD who are able to attend weekly clinic appointments
* Age 19-64, not pregnant and either sterile or using a medically acceptable method of birth control
* A willingness and ability to provide competent signed informed consent
* A level of understanding sufficient to perform all tests and examinations required by the protocol (including fluency of spoken English)

Exclusion Criteria:

* Any diagnosis of schizophrenia or bipolar I disorder, or active substance dependence
* Unstable general medical condition or serious illness (e.g.. death or hospitalization is anticipated within one year), poor kidney function, liver function (defined as lab values ≥ three times the upper limit of the laboratory normal) and seizure disorders with the exception of childhood seizure disorders.
* Subjects with prior non-response to Geodon for the treatment of PTSD with an adequate trial
* Enrollment in any study drug within the last 30 days. Current pharmacotherapy is permitted, provided that the medication and dose have been stable for the past 90 days.
* Pregnancy or nursing
* Any subject judged clinically to be at serious suicidal risk in the opinion of the investigator

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2002-12; Study Completion 2005-04

PRIMARY OUTCOMES:
Response to ziprasidone or placebo (inactive drug) will be measured by Clinician Administered PTSD Scale (CAPS) and Treatment Outcomes PTSD Scale (TOP-8).

SECONDARY OUTCOMES:
A secondary aim of the study is to measure effects on depression and anxiety symptoms in the same persons, using the HAM-A, HAM-D and the CGI. Quality of life will also be assessed using the QOLI.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Petty, MD, PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Psychiatry and Research Center, Omaha, Nebraska, United States